CLINICAL TRIAL: NCT01114490
Title: A Single Dose Study to Investigate the Pharmacokinetics of MK0859 in Patients With Hepatic Insufficiency
Brief Title: Pharmacokinetics of Anacetrapib (MK0859) in Patients With Hepatic Insufficiency (MK-0859-039)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0859-039; 2010_530
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Dyslipidemia
Keywords: Hepatic Insufficiency
MeSH Terms: conditions — Dyslipidemias; Hepatic Insufficiency | interventions — anacetrapib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1 - Group 1 (Experimental): Moderate Hepatic Patients
  Interventions: Drug: anacetrapib
- Part 1 - Group 2 (Experimental): Healthy Subjects
  Interventions: Drug: anacetrapib
- Part 2 - Group 1 (Experimental): Mild Hepatic Patients
  Interventions: Drug: anacetrapib
- Part 2 - Group 2 (Experimental): Healthy Subjects
  Interventions: Drug: anacetrapib

INTERVENTIONS:
Drug: anacetrapib — single dose administration of anacetrapib (MK0859) 100 mg oral tablet

SUMMARY:
This study will evaluate the Area Under the Curve (AUC(0 to infinity)) of anacetrapib.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of reproductive potential test negative for pregnancy and agree to use two acceptable methods of birth control throughout the study
* Subject is in good health
* Subject agrees to refrain from consumption of red wine, grapefruit, orange and apple juices throughout the study

Exclusion Criteria:

* Patient has a history of cancer
* Patient is a nursing mother
* Patient is unable to refrain from or anticipates the use of any prescription or non-prescription medication during the study
* Patient consumes excessive amounts of alcohol or caffeine
* Patient has had major surgery, donated blood or participated in another investigational study within the past 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC(0 to infinity)) of anacetrapib | through 168 hours post dose

SECONDARY OUTCOMES:
Tolerability of a single dose administration of 100mg anacetrapib, measured by the number of clinical and laboratory adverse events | through 14 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Lauring B, Li XS, Liu Y, Corr C, Lazarus N, Cote J, Larson P, Levonas AO, Lasseter KC, Preston RA, Smith WB, Lai E, Wagner JA. Influence of renal and hepatic impairment on the pharmacokinetics of anacetrapib. J Clin Pharmacol. 2014 Nov;54(11):1247-55. doi: 10.1002/jcph.320. Epub 2014 Jun 6. PMID 24782116